CLINICAL TRIAL: NCT00968994
Title: A Randomized, Site-Matched, Controlled Trial of exSALT SD7™ Compared to Xeroform® Petrolatum Dressing for the Management of Partial Thickness Donor Sites
Brief Title: Trial of exSALT SD7™ Compared to Xeroform® Petrolatum Dressing for the Management of Partial Thickness Donor Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Exciton Technologies Inc. (Industry)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Epidemiology Coordinating and Research Centre, Canada (Other); Smart Medical Research Inc. (Industry)
Responsible Party: Mr. Rod Precht / President & COO, Exciton Technologies Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-0004
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Wound Healing; Wound Infection
Keywords: Wound Healing; Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exSALT SD7™ Wound Dressing (Experimental): The exSALT™ SD7 Wound Dressing provides an antimicrobial barrier that inhibits microbial growth in the dressing. The exSALT™ SD7 Wound Dressing consists of 3 layers: two non-adherent polyethylene mesh wound contact layers and one absorbent core made of polyester. All three layers are silver coated. The concentration of silver on the exSALT™ SD7 Wound Dressing is approximately 0.4 mg/cm2 (2.5% w/w).
  Interventions: Device: The exSALT™ SD7 Wound Dressing
- Xeroform® Petrolatum Dressing (Active Comparator): Xeroform® Petrolatum Dressing (Xeroform® / Control Dressing) is fine mesh gauze impregnated with 3% Bismuth Tribromophenate in a special petrolatum blend. The dressing is a non adherent dressing that clings and conforms to all body parts.
  Interventions: Device: Xeroform® Petrolatum Dressing

INTERVENTIONS:
Device: The exSALT™ SD7 Wound Dressing — The exSALT™ SD7 Wound Dressing is indicated for the management of partial and full thickness wounds, including decubitus ulcers, venous stasis ulcers, diabetic ulcers, first and second degree burns, grafts and donor sites, or other acute or chronic wounds. The dressing may be used over debrided and grafted wounds.
  Other Names: K083870
  Arms: exSALT SD7™ Wound Dressing
Device: Xeroform® Petrolatum Dressing — Sterile, single use, non-adherent dressing consisting of absorbent gauze impregnated with Xeroform in a petrolatum blend.
  Other Names: K973507
  Arms: Xeroform® Petrolatum Dressing

SUMMARY:
This randomized, controlled trial is designed to evaluate split-thickness donor sites treated with exSALT SD7™ compared to donor sites treated with Xeroform®. For the purpose of this study, subjects enrolled will have selected donor sites or portions of donor sites designated as "Test Sites." The selected locations will be randomly assigned treatment with either the Test Dressing or the Control Dressing.

The primary objective of the trial will be to quantify the proportion of the donor sites in each group that are healed at 10 and 14 days. Secondary objectives will include: time to re-epithelialization, pain with dressing changes and mobilization, ease of use, resource utilization and safety, as well as quality of healing and overall cosmetic result. A total of 25 subjects will be enrolled in the trial.

The trial duration will be 12 weeks. For the purposes of this trial, healing will be defined as ≥ 90% re-epithelialization and must be visually confirmed by the investigator or designate and two other people (i.e., research nurse, burn resident, member of the Wound Care Team). The maximum time to evaluate healing will be 14 days +/-2 days. A final visit will be conducted at 12 weeks for safety and to evaluate the quality of healing.

DETAILED DESCRIPTION:
Autologous skin grafting is a common procedure required in the care of burn and plastic surgery patients where the harvesting of autologous skin grafts results in the creation of a partial thickness wound known as a donor site. The donor site healing time can affect the length of hospitalization and subject survival.

The literature reports the use of a variety of donor site dressing materials including fine mesh gauze, polyurethane film, synthetic fiber and hydrocolloids (Kilinc, Sensoz et al. 2001). The literature reports what might be considered the optimal donor site dressing attributes. These attributes would include: minimizing pain, velocity in healing, minimizing bacterial growth and simplicity in use (Rakel, Bermel et al. 1998).

However, none of the available dressing products are entirely satisfactory. Fine mesh gauze (FMG) is the donor site dressing used at many burn centers, as it is inexpensive, can be placed on posterior donor sites, does not require a margin of intact skin and allows large amounts of exudate to drain away from the donor site.

However, FMG does not have any inherent anti-infective properties and provides a dry environment for wound healing. Xeroform® Petrolatum Dressing resembles FMG physically except that it contains 3% xeroform (bismuth tribromophenate) which exerts some antibacterial effect (Feldman, Rogers et al. 1991). Xeroform® Petrolatum Dressing is the standard donor site dressing in the Firefighters' Burn Treatment Unit (3C2 WMC) and Plastic Surgery Unit (3D3 WMC) and has been selected as the control treatment (Control Dressing).

Research evidence demonstrates that partial thickness wounds re-epithelialize more rapidly in a moist environment that is free from infection (Alper 1986; Alvarez 1988). In an effort to provide an improved method of dressing wounds and donor sites, exSALT SD7™ has been proposed as an alternative dressing (Test Dressing). The dressing is intended to reduce pain and discomfort and improve the re-epithelialization process by providing a moist environment. The model outlined in this protocol provides the basis for a controlled comparison of wound healing and re-epithelialization in a clean partial thickness wound that allows us to compare the healing rate and quality of the Test Dressing compared to our standard of care to determine safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* signed or verbal informed consent provided
* are 18 to 65 years of age
* scheduled to undergo a split-thickness skin graft (autograft) that will result in a donor site or sites that are; a first time harvest and includes primarily the anterior including medial and lateral aspects of the anterior portion(s) of the thigh(s) with either; a single donor site that is a minimum of 8 x 20 cm or two donor sites are both a minimum of 8 x 8 cm and the resulting test sites are generally comparable in size and wound characteristics.
* requires hospitalization for initial treatment

Exclusion Criteria:

* require full thickness graft
* known skin sensitivity to any of the dressing components
* poor prognosis and who are unlikely to survive the trial period
* participating in another concurrent trial
* exhibiting any other medical condition, which, according to the investigator, justifies the subject's exclusion from the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the proportion of donor sites healed. | 10 days
Evaluate the proportion of donor sites healed. | 14 Days

SECONDARY OUTCOMES:
Time to re-epithelialization. | 12 weeks
Pain with dressing changes and mobilization. | 12 weeks
Assessments that quantify ease of use. | 12 weeks
Resource utilization and safety. | 12 weeks
Appearance and long term cosmetic results. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Collins-Nakai, MD, MBA, Study Director — Exciton Technologies Inc.; Edward E Tredget, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- The University of Alberta Hospital, Edmonton, Alberta, Canada